CLINICAL TRIAL: NCT04657692
Title: Incidence of Complications Associated With Anesthesia in Obesity Parturient Undergoing Cesarean Delivery- a Retrospective Review
Brief Title: Incidence of Complications Associated With Anesthesia in Obesity Parturient Undergoing Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 873/2562 (EC2); Si 125/2020 (Other: Siriraj Institutional Review Board)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Cesarean Section Complications; Anesthesia Complication; Obesity, Morbid
Keywords: anesthetic complications; maternal outcomes; neonatal outcomes; cesarean section; obesity
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Anesthesia; Amino Acid Motifs

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Anesthesia; general or regional — General anesthesia: general anesthesia with endotracheal tube Regional anesthesia: spinal anesthesia, epidural anesthesia, combined spinal epidural anesthesia

SUMMARY:
The incidence of obesity parturient has been increasing worldwide. There was a report revealing one third of pregnant women in United state considered obesity.

Obesity is associated with increased in maternal and neonatal complications. Also, there was an increasing in the rate of cesarean delivery. Anesthetic management of the obese parturient is differ from non-obese parturients. There were higher risk of difficult intubation, failed intubation, pulmonary aspiration and difficult regional anesthesia such as spinal anesthesia or epidural catheter placement comparing with non-obese parturient.

The aim of the study is to report complication associated with anesthesia in obese patients undergoing cesarean delivery in Single University hospital, Bangkok, THAILAND.

DETAILED DESCRIPTION:
The incidence of obesity parturient has been increasing worldwide. There was a report revealing one third of pregnant women in United state considered obesity.

Obesity is associated with increased in maternal and neonatal complications. Also, there was an increasing in the rate of cesarean delivery. Anesthetic management of the obese parturient is differ from non-obese parturients. There were higher risk of difficult intubation and difficult regional anesthesia such as spinal anesthesia or epidural catheter placement comparing with non-obese parturient.

WHO categorised obesity into 3 classification; grade 1: BMI 30-34.9 kg/m2, grade 2: BMI 35-39.9 kg/m2, grade 3: BMI > 40 kg/m2. This study emphasised in grade 3 obese pregnant women (BMI>40 kg/m2) undergoing cesarean delivery that were at risk of increasing in anesthetic complications such as airway complications as well as complications derived from regional anesthesia eg. high spinal block, failed spinal block etc.

Therefore, the primary objective of the study is to report complication associated with anesthesia in obese patients undergoing cesarean delivery in Single University hospital, Bangkok, THAILAND. The secondary objectives rate of postpartum haemorrhage, rate of hysterectomy and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women BMI>,= 40 kg/m2 underwent cesarean delivery

Exclusion Criteria:

* Patients with gestational age <,= 24 weeks
* Patients with death fetus in Utero
* Multiple gestation
* Patients with intrapelvic cavity pathology eg. myoma uteri
* Patients with abnormal placentation
* Patients with polyhydramnios

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese pregnant women whose body mass index (BMI>,= 40 kg/m2) underwent cesarean delivery
Sampling Method: Non-Probability Sample
Enrollment: 527 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of complications | intraoperative period to 24 hours postoperative
  Incidence of maternal complications associated with anesthesia

SECONDARY OUTCOMES:
Incidence of obstetric-related complications | intraoperative period to 24 hours postoperative
  Incidence of maternal complicaitions associated with obstetrics eg. amount of hemorrhage, rate of hysterectomy, rate of blood transfusion
Neonatal outcomes | Neonate apgar score at 1-min and 5 min
  Neonate apgar score (ranging 0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Patchareya Nivatpumin, M.D., Principal Investigator — Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Patchareya Nivatpumin, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nivatpumin P, Lertbunnaphong T, Maneewan S, Vittayaprechapon N. Comparison of perioperative outcomes and anesthetic-related complications of morbidly obese and super-obese parturients delivering by cesarean section. Ann Med. 2023 Dec;55(1):1037-1046. doi: 10.1080/07853890.2023.2187877. PMID 36947155